CLINICAL TRIAL: NCT04196452
Title: Long-term Follow-up of Ipilimumab-treated Pediatric Patients Enrolled in the Dutch Melanoma Treatment Registry (DMTR)
Brief Title: A Retrospective Observational Study on the Long-term Effects of Ipilimumab-treated Pediatric Participants in the Dutch Melanoma Treatment Registry (DMTR)
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-557
Record Dates: First submitted 2019-12-11; First posted 2019-12-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: participants 12 to under 18
  Interventions: Drug: Ipilimumab
- Arm B: participants under 12
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Specified dose on specified days

SUMMARY:
This is an observational, national, retrospective study consisting of pediatric patients with advanced (spread or unremoveable) melanoma identified in the DMTR in the Netherlands

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trials, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Less than 18 years of age at first dose of monotherapy Ipilimumab used for treatment of advanced melanoma
* Histological or cytological confirmation of advanced (unresectable or metastatic) melanoma

Exclusion Criteria:

-Participation in a clinical trial within the past 4 weeks prior to first dose with ipilimumab or concurrently

Other inclusion/exclusion criteria apply

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes participants who are under 18 years old who are diagnosed with advanced (unresectable or metastatic) melanoma who have been treated with ipilimumab and enrolled in the DMTR
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2034-02-20 (Estimated); Study Completion 2034-07-24 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) Grades 3-4 | up to 10 years

SECONDARY OUTCOMES:
Baseline assessment of population demographics | up to 10 years
Baseline assessment of comorbidities | up to 10 years
Baseline assessment of disease characteristics | up to 10 years
Baseline assessment of treatment history | up to 10 years
Assessment of ipilimumab dose exposure | up to 10 years
Assessment of changes in ipilumamb treatment: dose interruptions/discontinuations | up to 10 years
Assessment of Ipilimumab dose frequency | up to 10 years
Assessment of ipilimumab treatment duration | up to 10 years
Assessment of ipilimumab number of infusions | up to 10 years
Overall Survival (OS) | up to 10 years
Time to progression (TTP) | up to 10 years
Assessment of physical growth and development | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html